CLINICAL TRIAL: NCT00929292
Title: Study of Growth and Gastrointestinal Tolerance of an Alpha-Lactalbumin Enriched and Probiotic-Supplemented Infant Formula in Infants With Colic.
Brief Title: Safety and Tolerance Study of Alpha-Lactalbumin Enriched and Probiotic-Supplemented Infant Formula in Infants With Colic
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sodilac (Industry)
Responsible Party: Pr Christophe Dupont, Hôpital Saint Vincent de Paul
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: DAH-CL3-001
Record Dates: First submitted 2009-06-26; First posted 2009-06-29 (Estimated); Last update posted 2009-06-29 (Estimated); Status verified 2009-06

CONDITIONS: Growth; Colic
Keywords: Infant formula; Alpha-lactalbumin; Protein composition; Colic; Probiotics
MeSH Terms: conditions — Colic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Modilac Dahlia 1 (Experimental): Formula enriched with alpha-lactalbumin and containing a probiotic
  Interventions: Other: Modilac Dahlia 1
- Modilac 1 (Placebo Comparator): Regular milk
  Interventions: Other: Modilac 1

INTERVENTIONS:
Other: Modilac Dahlia 1 — Infant formula used for non breastfed children with colic
  Other Names: Dahlia
  Arms: Modilac Dahlia 1
Other: Modilac 1 — Infant formula used for non breastfed children
  Other Names: Modilac
  Arms: Modilac 1

SUMMARY:
The purpose of this study is to evaluate the nutritional adequacy, the digestive tolerance and the effect on colic of an alpha-lactalbumin-enriched and probiotic-supplemented infant formula.

DETAILED DESCRIPTION:
This double-blind, placebo-controlled study was undertaken with 66 healthy infants with colic, aged 3 weeks to 3 months, fed a month either with the experimental formula (EF) or with the control formula (CF) and evaluated for efficacy and safety parameters at days 15 and 30.

Both parents provided informed written consent.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term infants with a gestational age ranging from 37 to 42 weeks
* Non breastfed children
* Infants with normal growth
* Infants presenting colic defined as crying periods at least 3 hours per days, 3 days per weeks, for more than 3 weeks
* These crying periods could be associated with other digestive troubles(gas, abdominal distensions, regurgitations)
* Apgar score > 5 to 7 minutes

Exclusion Criteria:

* Infants with severe regurgitations
* Newborn currently participating in another trial
* Infants presenting a metabolic, nervous or organic disease able to interfere with the study
* Infants presenting lactose intolerance
* Evidence of protein cow's milk allergy
* Mother who wants to keep breasfeeding

Ages: 3 Weeks to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2006-11; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Crying duration per 24 hours | 1 day before the first consumption ; 3 days before days 15 and 30

SECONDARY OUTCOMES:
Growth Parameters | Day 30
Clinical Tolerance | 3 days before days 15 and 30
Number of therapeutic failures (no diminution in the intensity or the frequency of the digestive symptoms) | Durind the 15 first days of the diet and during the 15 last days of the diet
Number of regurgitations per day | 3 days before days 15 and 30
Gas and abdominal distensions | 3 days before days 15 and 30
Necessary Additive treatments | 3 days before days 15 and 30
Parents' satisfaction | Days 15 and 30
Agitation/Restlessness Period Duration | 3 days before days 15 and 30

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Dupont, PhD, Principal Investigator — Hôpital Saint Vincent de Paul
Locations (12):
- France (12):
  - Dr Francine Gressin-Cohen, Antony
  - Hôpital privé d'Antony, Antony
  - Hôpital Robert Ballanger, Aulnay-sous-Bois
  - Dr Brigitte Pacault, Boulogne-Billancourt
  - Dr Michel Dogneton, Boulogne-Billancourt
  - Dr Nassira Belaroussi Maamri, Boulogne-Billancourt
  - Dr KALINDJIAN, Issy-les-Moulineaux
  - Groupe Hospitalier de l'Institut Catholique de Lille (GHICL), Lille
  - Dr Christophe Grillon, Meaux
  - Dr COUPRIE Claire, Paris
  - Dr RONZIER Monique, Paris
  - Dr Locquet André, Roncq